CLINICAL TRIAL: NCT00721500
Title: An Evaluation of the Lens Fit of Narafilcon A Soft Contact Lenses
Brief Title: A Comparison of Two Daily Disposable Contact Lenses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-0812; PROD-502
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Results first posted 2011-03-02 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Refractive Error; Myopia
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- narafilcon A / etafilcon A - etafilcon A - narafilcon A (Experimental): First, narafilcon A and etafilcon A contact lenses worn contralaterally. Second, etafilcon A contact lenses worn in both eyes. Third, narafilcon A contact lenses worn in both eyes.
  Interventions: Device: etafilcon A; Device: narafilcon A
- narafilcon A / etafilcon A - narafilcon A - etafilcon A (Experimental): First, narafilcon A and etafilcon A contact lenses worn contralaterally. Second, narafilcon A contact lenses worn in both eyes. Third, etafilcon A contact lenses worn in both eyes.
  Interventions: Device: etafilcon A; Device: narafilcon A
- narafilcon A - etafilcon A - narafilcon A / etafilcon A (Experimental): First, narafilcon A contact lenses worn in both eyes. Second, etafilcon A contact lenses worn in both eyes. Third, narafilcon A and etafilcon A contact lenses worn contralaterally.
  Interventions: Device: etafilcon A; Device: narafilcon A
- etafilcon A - narafilcon A - narafilcon A / etafilcon A (Experimental): First, etafilcon A contact lenses worn in both eyes. Second, narafilcon A contact lenses worn in both eyes. Third, narafilcon A and etafilcon A contact lenses worn contralaterally.
  Interventions: Device: etafilcon A; Device: narafilcon A

INTERVENTIONS:
Device: etafilcon A — contact lens
  Other Names: 1-Day Acuvue Moist
Device: narafilcon A — contact lens
  Other Names: TruEye

SUMMARY:
This study seeks to evaluate the clinical fitting performance of a new daily disposable contact lens to an existing daily disposable contact lens.

ELIGIBILITY:
Inclusion Criteria:

* They are of legal age (18 years) and capacity to volunteer.
* They understand their rights as a research subject and are willing to sign a Statement of Informed Consent.
* They are willing and able to follow the protocol.
* They would be expected to attain at least 6/9 (20/30) in each eye with the study lenses.
* They are able to wear contact lenses with a back vertex power of -1.00 to -6.00DS.
* They have a maximum of 1.00D of refractive astigmatism (i.e. ≤ 1.00 DC).
* They have successfully worn contact lenses within six months of starting the study.

Exclusion Criteria:

* They have an ocular disorder which would normally contra-indicate contact lens wear.
* They have a systemic disorder which would normally contra-indicate contact lens wear.
* They are using any topical medication such as eye drops or ointment.
* They are aphakic.
* They have had corneal refractive surgery.
* They have any corneal distortion resulting from previous hard or rigid lens wear or has keratoconus.
* They are pregnant or lactating.
* They have grade 2 or greater of any of the following ocular surface signs: corneal oedema, corneal vascularisation, corneal staining, tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
* They have any infectious disease (e.g. hepatitis) or any immunosuppressive disease (e.g. HIV).
* They have diabetes.
* They have taken part in any other clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Visioncare Research Ltd, Farnham, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 25 subjects enrolled to the study.
Pre-assignment Details: Subjects were enrolled per inclusion/exclusion criteria and randomized to a study arm.
Groups:
- Narafilcon A/Etafilcon A - Etafilcon A - Narafilcon A: First, narafilcon A and etafilcon A contact lenses worn contralaterally. Second, etafilcon A contact lenses worn in both eyes. Third, narafilcon A contact lenses worn in both eyes.
- Narafilcon A/Etafilcon A - Narafilcon A - Etafilcon A: First, narafilcon A and etafilcon A contact lenses worn contralaterally. Second, narafilcon A contact lenses worn in both eyes. Third, etafilcon A contact lenses worn in both eyes.
- Narafilcon A - Etafilcon A - Narafilcon A/Etafilcon A: First, narafilcon A contact lenses worn in both eyes. Second, etafilcon A contact lenses worn in both eyes. Third, narafilcon A and etafilcon A contact lenses worn contralaterally.
- Etafilcon A - Narafilcon A - Narafilcon A/Etafilcon A: First, etafilcon A contact lenses worn in both eyes. Second, narafilcon A contact lenses worn in both eyes. Third, narafilcon A and etafilcon A contact lenses worn contralaterally.
Period: Period One
Arm/Group | Narafilcon A/Etafilcon A - Etafilcon A - Narafilcon A | Narafilcon A/Etafilcon A - Narafilcon A - Etafilcon A | Narafilcon A - Etafilcon A - Narafilcon A/Etafilcon A | Etafilcon A - Narafilcon A - Narafilcon A/Etafilcon A
Started | 6 | 7 | 6 | 6
Completed | 6 | 7 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period Two
Arm/Group | Narafilcon A/Etafilcon A - Etafilcon A - Narafilcon A | Narafilcon A/Etafilcon A - Narafilcon A - Etafilcon A | Narafilcon A - Etafilcon A - Narafilcon A/Etafilcon A | Etafilcon A - Narafilcon A - Narafilcon A/Etafilcon A
Started | 6 | 7 | 6 | 6
Completed | 6 | 7 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period Three
Arm/Group | Narafilcon A/Etafilcon A - Etafilcon A - Narafilcon A | Narafilcon A/Etafilcon A - Narafilcon A - Etafilcon A | Narafilcon A - Etafilcon A - Narafilcon A/Etafilcon A | Etafilcon A - Narafilcon A - Narafilcon A/Etafilcon A
Started | 6 | 7 | 6 | 6
Completed | 6 | 7 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled and completed subjects were included in the baseline summary.
Groups:
- All Subjects: All subjects who enrolled and completed study.
Arm/Group | All Subjects
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 8
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes Successfully Fit
Description: Overall lens fit acceptance was assessed by the Investigator based on lens fit alone in a 6-level scale; 0=should not be worn, 1=should not be dispensed although no immediate danger, 2=borderline but unacceptable, 3=minimal acceptable, early review, 4=not perfect but OK to dispense and 5=perfect. Lens fitting responses >2 were considered 'successful fit' while the rest of responses were considered 'unsuccessful fit'.
Time Frame: Within 20 minutes of lens insertion
Population: Participants who were enrolled and completed the study.
Measure: Number; unit: proportion of participant eyes
Units Other Than Participants: eyes
Groups:
- Narafilcon A (Bilateral): narafilcon A contact lens worn in both eyes.
- Narafilcon A (Contralateral): Narafilcon A worn in either eye.
- Etafilcon A (Bilateral): Etafilcon A contact lens worn in both eyes.
- Etafilcon A (Contralateral): Etafilcon A worn in either eye.
Arm/Group | Narafilcon A (Bilateral) | Narafilcon A (Contralateral) | Etafilcon A (Bilateral) | Etafilcon A (Contralateral)
Number analyzed (Participants) | 25 | 25 | 25 | 25
Number analyzed (eyes) | 50 | 25 | 50 | 25
proportion of participant eyes | 0.98 | 0.96 | 0.96 | 0.96

2. Primary Outcome: Lens Fit Decentration
Description: Lens centration was assessed in primary gaze, diffuse white light, low-medium magnification, with graticule. Lens fit decentration with respect to visible cornea was measured to nearest 0.1mm.
Time Frame: Within 20 minutes of lens insertion
Population: Participants who were enrolled and completed the study.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eye
Groups:
- Narafilcon A: Narafilcon A contact lens worn in both eyes.
Arm/Group | Narafilcon A | Narafilcon A (Contralateral) | Etafilcon A (Bilateral) | Etafilcon A (Contralateral)
Number analyzed (Participants) | 25 | 25 | 25 | 25
Number analyzed (eye) | 50 | 25 | 50 | 25
mm | 0.25 (0.14) | 0.22 (0.16) | 0.27 (0.17) | 0.27 (0.15)

3. Primary Outcome: Lens Tightness on Cornea With Manual Digit Push Up
Description: Lens tightness on push-up assessed by digital push-up test (gentle push of the lens upward using the lower lid) with eye in primary gaze position and observing ease of push-up and speed of return to original position. Tightness is measured on a 0%-100% continuous scale where 0%=falls from cornea without lid support, 50%=optimum and 100%=no movement.
Time Frame: Within 20 minutes of lens insertion
Population: Participants who were enrolled and completed the study.
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: eye
Arm/Group | Narafilcon A (Bilateral) | Narafilcon A (Contralateral) | Etafilcon A (Bilateral) | Etafilcon A (Contralateral)
Number analyzed (Participants) | 25 | 25 | 25 | 25
Number analyzed (eye) | 50 | 25 | 50 | 25
percentage | 44.6 (6.3) | 46.9 (5.5) | 56.3 (8.6) | 58.1 (7.8)

ADVERSE EVENTS:
Arm/Group | Narafilcon A/Etafilcon A - Etafilcon A - Narafilcon A | Narafilcon A/Etafilcon A - Narafilcon A - Etafilcon A | Narafilcon A - Etafilcon A - Narafilcon A/Etafilcon A | Etafilcon A - Narafilcon A - Narafilcon A/Etafilcon A
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.